CLINICAL TRIAL: NCT02733445
Title: Assessment of Metabolic Outcomes Among Patients With Chronic Myelogenous Leukemia (CML) Initiating Therapy With a Tyrosine Kinase Inhibitor (TKI)
Brief Title: Metabolic Outcomes in Patients Receiving Tyrosine Kinase Inhibitor (TKI) Therapy With Dasatinib or Nilotinib
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA180-633
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Myeloid Leukemia (CML)
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib; nilotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- dasatinib cohort: Patients with CML receiving dasatinib
  Interventions: Drug: dasatinib
- nilotinib cohort: Patients with CML receiving nilotinib
  Interventions: Drug: nilotinib

INTERVENTIONS:
Drug: dasatinib
  Groups: dasatinib cohort
Drug: nilotinib
  Groups: nilotinib cohort

SUMMARY:
The purpose of this study was to determine how often and how likely patients are to develop Type 2 Diabetes or high cholesterol/lipids when receiving dasatinib or nilotinib as therapy for Chronic Myelogenous Leukemia (CML).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* At least 1 prescription for nilotinib or dasatinib between 7/1/2006-12/31/2014
* Continuously enrolled in the same health plan throughout the study period
* At least 2 diagnosis codes for CML at least 30 days apart as documented in medical insurance claims

Exclusion Criteria:

* patients who had a documented diagnosis of diabetes in their medical claims or received a medication for diabetes before receiving dasatinib or nilotinib
* patients who had a documented diagnosis of high cholesterol/lipids in their medical claims or received a medication for high cholesterol/lipids before receiving dasatinib or nilotinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study is based on health insurance claims data, which covers inpatient and outpatient claims from a geographically diverse area across the U.S.
Sampling Method: Non-Probability Sample
Enrollment: 2650 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
incidence rate of new-onset Type 2 Diabetes (T2DM) among patients with Chronic myelogenous leukemia (CML) receiving imatinib as first-line therapy in a commercially or Medicare insured population | approximately 101 months
incidence rate of new-onset Type 2 Diabetes (T2DM) among patients with Chronic myelogenous leukemia (CML) receiving dasatinib as first-line therapy in a commercially or Medicare insured population | approximately 101 months
incidence rate of new-onset Type 2 Diabetes (T2DM) among patients with Chronic myelogenous leukemia (CML) receiving nilotinib as first-line therapy in a commercially or Medicare insured population | approximately 101 months
incidence rate of new-onset Hyperlipidemia (HLD) among patients with Chronic myelogenous leukemia (CML) receiving imatinib as first-line therapy in a commercially or Medicare insured population | approximately 101 months
incidence rate of new-onset Hyperlipidemia (HLD) among patients with Chronic myelogenous leukemia (CML) receiving dasatinib as first-line therapy in a commercially or Medicare insured population | approximately 101 months
incidence rate of new-onset Hyperlipidemia (HLD) among patients with Chronic myelogenous leukemia (CML) receiving nilotinib as first-line therapy in a commercially or Medicare insured population | approximately 101 months

SECONDARY OUTCOMES:
incidence rate of new-onset Type 2 Diabetes (T2DM) among patients with Chronic myelogenous leukemia (CML) receiving dasatinib as first- or second-line therapy in a commercially or Medicare insured population | approximately 101 months
incidence rate of new-onset Type 2 Diabetes (T2DM) among patients with Chronic myelogenous leukemia (CML) receiving nilotinib as first- or second-line therapy in a commercially or Medicare insured population | approximately 101 months
incidence rate of new-onset Hyperlipidemia (HLD) among patients with Chronic myelogenous leukemia (CML) receiving dasatinib as first- or second-line therapy in a commercially or Medicare insured population | approximately 101 months
incidence rate of new-onset Hyperlipidemia (HLD) among patients with Chronic myelogenous leukemia (CML) receiving nilotinib as first- or second-line therapy in a commercially or Medicare insured population | approximately 101 months
risk comparison of developing Type 2 Diabetes (T2DM) among patients treated with imatinib with respect to patients treated with dasatinib as first-line therapy and as first- or second-line therapy | approximately 101 months
risk comparison of developing Type 2 Diabetes (T2DM) among patients treated with nilotinib with respect to patients treated with dasatinib as first-line therapy and as first- or second-line therapy | approximately 101 months
risk comparison of developing Hyperlipidemia (HLD) among patients treated with imatinib with respect to patients treated with dasatinib as first-line therapy and as first- or second-line therapy | approximately 101 months
risk comparison of developing Hyperlipidemia (HLD) among patients treated with nilotinib with respect to patients treated with dasatinib as first-line therapy and as first- or second-line therapy | approximately 101 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx